CLINICAL TRIAL: NCT00714207
Title: Evaluation of Adolescent Smoking Cessation Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Truth Initiative (Other)
Responsible Party: Alain Joffe, MD, MPH, Principal Investigator, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.32.01.12.04.A1
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Smoking Status
Keywords: adolescents; smoking; smoking cessation; tobacco use
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NOT Intervention (Experimental): Students in this arm of the study were randomized to receive the reformatted NOT program
  Interventions: Behavioral: NOT program
- NOT controls (Active Comparator): Students in this arm were randomized to receive a single group session on smoking cessation and were given youth oriented informational pamphlets on smoking cessation
  Interventions: Behavioral: NOT controls
- KB intervention (Experimental): Students in this arm of the study were randomized to receive the reformatted Kicking Butts intervention
  Interventions: Behavioral: Kicking Butts intervention
- KB controls (Active Comparator): Students in this arm were randomized to receive a single group session on smoking cessation and were given youth oriented informational pamphlets on smoking cessation
  Interventions: Behavioral: KB controls

INTERVENTIONS:
Behavioral: NOT program — Students in this arm of the study received the reformatted NOT intervention
  Arms: NOT Intervention
Behavioral: NOT controls — Students in this arm were randomized to receive a single group session on smoking cessation and were given youth oriented informational pamphlets
  Arms: NOT controls
Behavioral: Kicking Butts intervention — Students in this arm of the study were randomized to receive the reformatted Kicking Butts intervention
  Arms: KB intervention
Behavioral: KB controls — Students in this arm were randomized to receive a single group session on smoking cessation and were given youth oriented informational pamphlets
  Arms: KB controls

SUMMARY:
The purpose of this study was to determine if a school-based multi-session group smoking cessation program is more effective than a single session group program.

DETAILED DESCRIPTION:
The investigators reformatted two group smoking cessation programs (the NOT program of the American Lung Association and Kicking Butts), both of which involve 50 minute sessions delivered once weekly, into a program that could be delivered during school lunch periods (25-30 minutes) twice weekly. Smoking status was subsequently assessed over the 12 month period following the intervention,

ELIGIBILITY:
Inclusion Criteria:

* Students who indicated they smoked cigarettes and wanted to quit

Exclusion Criteria:

* Students referred as part of a disciplinary requirement to stop smoking

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 407 (Actual)
Dates: Start 2002-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Self reported quit status (Student identifies self as non-smoker and no smoking for 30 days) | End of program and 1, 3, 6 and 12 months later

SECONDARY OUTCOMES:
Salivary cotinine level | End of program and 1, 6 and 12 months later

CONTACTS AND LOCATIONS:
Overall Officials: Alain Joffe, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (8):
- United States (8):
  - Northwestern High School, Baltimore, Maryland
  - Walbrook High School, Baltimore, Maryland
  - Patterson High School, Baltimore, Maryland
  - Southern High School/Digital Harbor, Baltimore, Maryland
  - Long Reach High School, Columbia, Maryland
  - Hammond High School, Columbia, Maryland
  - Mount Hebron High School, Ellicott City, Maryland
  - Howard High School, Ellicott City, Maryland

REFERENCES:
- [Derived] Joffe A, McNeely C, Colantuoni E, An MW, Wang W, Scharfstein D. Evaluation of school-based smoking-cessation interventions for self-described adolescent smokers. Pediatrics. 2009 Aug;124(2):e187-94. doi: 10.1542/peds.2008-2509. Epub 2009 Jul 27. PMID 19651564